CLINICAL TRIAL: NCT06476483
Title: Implementing the DIALOG Outcome Measure and a Solution-Focused Intervention (DIALOG+) in a Rehabilitation Psychiatric Inpatient Setting: A Mixed Methods Feasibility Study
Brief Title: Feasibility and Acceptability of Implementing DIALOG+ in a Psychiatric Rehabilitation Unit
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 187799
Record Dates: First submitted 2024-05-20; First posted 2024-06-26 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-05

CONDITIONS: Psychological Recovery

STUDY DESIGN:
Intervention Model Description: Feasibility and acceptability study.
  A mixed methods design will be used to meet the aims of this study. The study will consist of two parts, firstly quantitative; quasi-experimental group comparison design and secondly a qualitative design with data collection based on focus groups and additional surveys being distributed to patients who participate.
  The independent variable will be membership of the comparison (DIALOG) or treatment (DIALOG+) group. The dependent variable will be scores on the DIALOG measure at the end of the intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DIALOG (Other): This is the comparison group, they will complete the DIALOG measure biweekly for 5 months. DIALOG scores pre and post-intervention will be used in the analyses.
  Interventions: Behavioral: DIALOG
- DIALOG+ (Active Comparator): This is the treatment group. The participants in this group have agreed to participate in DIALOG+ and will receive the intervention biweekly for 10 sessions (5 months). Pre and post-intervention DIALOG scores will be used in the analysis.
  Interventions: Behavioral: DIALOG+

INTERVENTIONS:
Behavioral: DIALOG+ — A person-centred and solution-focused intervention linked to the DIALOG outcome measure (a measure of patient experience and quality of life).
  Arms: DIALOG+
Behavioral: DIALOG — An outcome measure consisting of 11 questions, with 8 related to quality of life and 3 items on treatment satisfaction. Patients can rate their satisfaction on a 7-point scale for each of the 8 life domains and 3 treatment aspects, resulting in scores for both quality of life and treatment satisfaction. The DIALOG scale does not provide any guidance for patient and clinician interactions.
  Arms: DIALOG

SUMMARY:
This study aims to understand if implementing DIALOG+ in an inpatient psychiatric rehabilitation setting is feasible (can the intervention be implemented) and acceptable (how the intervention is perceived by staff and patient participants). If the intervention is proven to be feasible and acceptable a larger-scale study may take place. This study has been developed in response to the trust-wide implementation of DIALOG outcome measures. DIALOG+ offers additional solution-focused and person-centred follow-up questions to the DIALOG questions and links to multidisciplinary team (MDT) discussions. It is hoped that the conversations had during DIALOG+ meetings will support positive outcomes, and the learning gathered from this study will drive change and improvement for other people requiring psychiatric rehabilitation inpatient admissions in the future. DIALOG+ has been successfully implemented in community settings in the national health service (NHS) but has not been implemented in psychiatric rehabilitation inpatient settings. This study will aim to recruit patient and staff participants from NHS psychiatric rehabilitation inpatient wards. Patient participants who will be eligible to take part are those who can consent, are between the ages of 18-65, and can complete DIALOG and DIALOG+. To understand the feasibility of the intervention, descriptive statistics will be collected and to understand acceptability focus groups will take place and surveys will be collected. Quantitative data collection will take place over 5 months and will be split into 2 groups. Group one will be a comparison group where participants will act as an extended baseline group and biweekly DIALOG outcomes will be collected. Group 2 will be a Treatment group and participants will receive the DIALOG+ intervention intervention, DIALOG outcomes will be collected biweekly as part of the intervention. Finally, there will be a period to gather qualitative feedback from patient participants using surveys, and from staff participants using focus groups or semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65
* Capacity to give informed consent as determined by the MDT and through following informed consent processes.
* Admitted into the inpatient ward
* Can complete DIALOG and DIALOG+

Exclusion Criteria:

* No capacity to consent
* Insufficient command of the English language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcome- Recruitment rate/consent rate | assessed at the end of the study (after 5 months)
  The number of people who agreed and consented to participate in the study out of the total number of eligible participants approached. Reported as a percentage.
Feasibility outcome- Number of eligible participants. | assessed at the end of the study (after 5 months)
  Eligible participants are those who meet the inclusion criteria, reported as a count of participants.
Feasibility outcome- Participation rate | assessed at the end of the study (after 5 months)
  The proportion of those who consented and agreed to engage in DIALOG and DIALOG+ out of the number of participants who engaged in the intervention after consenting. Reported as a percentage of participants.
Feasibility outcome- Completion rate | assessed at the end of the study (after 5 months)
  The proportion of those who completed the intervention out of the number who consented and engaged in DIALOG and DIALOG+. Reported as a percentage of participants.
Feasibility outcome- Drop out rate | assessed at the end of the study (after 5 months)
  The number of participants who completed the intervention out of total number of patients enrolled. Reported as a percentage of participants.
Feasibility outcomes- Reasons for drop out | assessed at the end of the study (after 5 months)
  Reasons for drop out will be assessed when by asking the participant after drop out.
Feasibility outcomes- Follow up rate | assessed at the end of the study (after 5 months)
  The number of patients willing to engage in follow-up surveys related to the study out of the total number of participants enrolled in the study. Reported as a percentage of participants.
Feasibility outcome- The willingness of clinicians to recruit participants | assessed at the end of the study (after 5 months)
  Number of staff members who attend DIALOG+ training and implement intervention out of the total number of staff offered to participate. Reported as a percentage.
Feasibility outcome- Average number of DIALOG+ sessions | assessed at the end of the study (5 months)
  Reported as the average number of participants.
Acceptability outcome- Cost | assessed at the end of the study (after 5 months)
  Analysing the cost and benefits of implementing the intervention (including staff training). Reported as a total amount or duration of time spent on training (minutes).
Number of staff participants who find DIALOG and DIALOG+ feasible and acceptable to implement in an inpatient rehabilitation setting. Assessed using thematic analysis of focus groups. | assessed at the end of the study (after 5 months)
  To assess the acceptability of the intervention a theoretical framework (Sekhon et al., 2017) was used. Feasibility objectives are defined by Bugge et al., 2013. Focus group transcripts will be subject to a qualitative thematic analysis. Analysis of focus groups will involve coding, organising coding into themes, reviewing themes, and generating a final thematic overview with in relation to the research question (Braun & Clarke, 2006).
Number of patients who find it feasible and acceptable to implement DIALOG and DIALOG+ in an inpatient rehabilitation setting. Assessed using thematic analysis and average scores of patient surveys. | assessed at the end of the study (after 5 months)
  The questionnaires will be a mixture of open ended questions and Likert Scale questions based on questions asked by Matanov et al. (2021), 8 of the questions are scored on a Likert scale (1-5). The survey will be given to patients post-intervention. Questions on the scale have been specifically developed to assess feasibility and acceptability of DIALOG+. An average total score will be used in the analysis of Likert scale questions. Open-ended questionnaire responses will be subject to a qualitative thematic analysis. Analysis will involve coding, organising coding into themes, reviewing themes, and generating a final thematic overview in relation to the research question (Braun & Clarke, 2006).

SECONDARY OUTCOMES:
DIALOG questionnaire | At the beginning of the study, then biweekly for a duration of 5 months with the final measure taken after 5 months
  The DIALOG questionnaire consists of 11 questions, with 8 items related to subjective quality of life (SQOL) and 3 items on treatment satisfaction. Patients can rate their satisfaction on a 7-point scale for each of the 8 life domains and 3 treatment aspects, resulting in scores for both SQOL and treatment satisfaction. An increase in score indicates improvement.
  The dependent variable will be DIALOG outcomes at the end of intervention or discharge and the independent variable will be the group binary variable (intervention or comparison group). Data will be analysed using a linear regression model to assess whether implementing DIALOG+ as an intervention in addition to using the DIALOG outcome measure, leads to improved outcomes.
  The unit of measure: reported as an average total score.
Demographic information | assessed at the end of the study (5 months)
  To gather demographic details from patients to assess the potential generalisability of DIALOG and DIALOG+. • Demographic information includes age, gender, ethnicity, history of mental illness or previous inpatient admissions, drug-use, diagnosis, baseline severity on DIALOG, and length of stay. Reported as a percentage of participants.
Length of admission in months | assessed at the end of the study (5 months)
  To use regression analysis to understand the effectiveness of the intervention and impact on admission length and DIALOG score.

CONTACTS AND LOCATIONS:
Locations (1):
- Forest Close, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data may be made openly available through the data repository at the University of Sheffield depending on the data sharing agreement with the Sheffield health and social care (SHSC).